CLINICAL TRIAL: NCT02584075
Title: Evaluate the Effect of Exenatide Treatment on Coronary Artery Endothelial Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Guang Wang, Director,Head of Endocrinology,Principal Investigator, Clinical Professor, Beijing Chao Yang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Exen100
Record Dates: First submitted 2015-10-15; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Coronary Endothelial Function
MeSH Terms: interventions — Exenatide; Metformin

ARMS (1):
- Lifestyle intervention (Experimental)
  Interventions: Drug: Byetta (Exenatide); Drug: Glucophage ( Metformin Hydrochloride)

INTERVENTIONS:
Drug: Byetta (Exenatide) — Exenatide treatment: 5 µg twice/day subcutaneous injection for 4 weeks, 10 µg twice/day subcutaneous injection for 8 weeks.
Drug: Glucophage ( Metformin Hydrochloride) — Metformin 500mg Tid

SUMMARY:
Type 2 diabetes mellitus (T2DM) is an important risk factor of cardio-cerebral vascular disease such as coronary heart disease. GLP-1 is a kind of incretin secreted by the L-cell located in Ileum. It acts as an incretin hormone by protentiating glucose-stimulated insulin release. Recent studies reported that GLP-1 RA can protect the vascular endothelial and prevent vascular from atherosclerosis. Investigators design this study to investigate exenatide's effect on the improvement of the coronary endothelial function by evaluating endothelium dependent diastolic function and testing the vascular endothelial active substance and related inflammatory factors.

ELIGIBILITY:
Inclusion Criteria:

* Females or males, and aged 20 to 65 years
* Newly diagnose type 2 diabetes mellitus with BMI>25kg/m2.
* HbA1C>8%.

Exclusion Criteria:

* Type 1 diabetes mellitus, diabetic ketoacidosis, diabetic hyperosmolar coma.
* Hepatic insufficiency (ALT or AST> 1.5*ULN).
* Renal insufficiency [Creatinine clearance rate (Ccr)]<60ml/min estimated from MDRD equation).
* Thyroid disease
* Use of any anti-diabetic, anti-hypertension or anti-dyslipidemia drugs.
* Pregnant or lactating woman.
* Severe anemia.
* Acute myocardial infarction or stoke.
* Other conditions at investigator's discretion.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Coronary endothelial function | the change of coronary endothelial function(baseline, 12 weeks)
  the change of coronary flow velocity reserve (CFVR)(baseline, 12 weeks)

SECONDARY OUTCOMES:
the changes of fasting plasma glucose (FPG) | the changes of fasting plasma glucose (FPG)(baseline, 12 weeks)
  the changes of fasting plasma glucose (FPG) (baseline, 12 weeks)
the changes of HbA1C | the changes of HbA1C(baseline, 12 weeks)
  the changes of HbA1C (baseline, 12 weeks)
the changes of fasting serum insulin (FINS) | the changes of fasting serum insulin (FINS) (baseline, 12 weeks)
  the changes of fasting serum insulin (FINS) (baseline, 12 weeks)
the changes of IL-1B | the changes of IL-1B (baseline, 12 weeks)
  the changes of IL-1B (baseline, 12 weeks)
the changes of IL-6 | the changes of IL-6 (baseline, 12 weeks)
  the changes of IL-6 (baseline, 12 weeks)
the changes of TNF-α | the changes of TNF-α(baseline, 12 weeks)
  the changes of TNF-α(baseline, 12 weeks)